CLINICAL TRIAL: NCT07078747
Title: Comparison of Video- and Model-Based Training in Developing Leopold Maneuver Skills Among Midwifery Students: A Randomized Controlled Trial
Brief Title: Video vs Model Training for Leopold Maneuver Skills
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kahramanmaras Sutcu Imam University (Other)
Responsible Party: Principal Investigator, Deniz Akyıldız, Assoc. Prof., Kahramanmaras Sutcu Imam University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Leopold Training
Record Dates: First submitted 2025-07-12; First posted 2025-07-22 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Midwifery Education; Clinical Skills Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Model-Based Training Group (Experimental): Participants in this group will receive the same 2-hour theoretical education, followed by hands-on practice of Leopold maneuvers on anatomical models under researcher supervision.
  Interventions: Behavioral: To compare the effectiveness of video- and model-based training methods in improving Leopold maneuver skills among midwifery students.
- Video-Based Training Group (Experimental): Participants in this group will receive a 2-hour theoretical education on Leopold maneuvers followed by video-based training using an instructional video. Training is conducted in a skills lab environment.
  Interventions: Behavioral: To compare the effectiveness of video- and model-based training methods in improving Leopold maneuver skills among midwifery students.
- Control Group (No Intervention): Participants in this group will only receive the 2-hour theoretical training. No additional practical training will be provided.

INTERVENTIONS:
Behavioral: To compare the effectiveness of video- and model-based training methods in improving Leopold maneuver skills among midwifery students. — This study involves two educational interventions aimed at improving Leopold maneuver skills among midwifery students. Both intervention groups receive a standardized 2-hour theoretical lecture about the purpose, application, and clinical relevance of the Leopold maneuvers.
  In the Video-Based Training Group, students watch an instructional video developed by the research team that visually demonstrates each step of the maneuver.
  In the Model-Based Training Group, students perform the maneuvers on anatomical models under the supervision of an instructor.
  These interventions are conducted in separate sessions to prevent cross-group contamination.
  Arms: Model-Based Training Group; Video-Based Training Group

SUMMARY:
This randomized controlled study aims to compare the effectiveness of video-based and model-based training methods in improving Leopold maneuver skills among second-year midwifery students. The study will be conducted at the Faculty of Health Sciences, Kahramanmaraş Sütçü Imam University. Eligible students will be randomly assigned into three groups: video-supported training, model-supported training, and control. All participants will first receive a 2-hour theoretical training session. Then, the video group will watch an instructional video, the model group will perform hands-on practice using anatomical models, and the control group will receive no additional intervention. Skill acquisition will be evaluated through practical assessments conducted a few days and two months after training. At the end of the study, compensatory training will be provided to all groups to ensure educational equity. Data collection tools include a psychomotor skills assessment form, a student satisfaction scale, and the Spielberger State Anxiety Inventory. Statistical analyses will be performed using SPSS software.

DETAILED DESCRIPTION:
This randomized controlled trial investigates the comparative effectiveness of video-based and model-based educational interventions in enhancing second-year midwifery students' psychomotor skills related to the Leopold maneuvers. The study is designed with three parallel arms: (1) video-supported training, (2) anatomical model-supported training, and (3) control (no additional intervention beyond theoretical instruction).

A total of eligible participants will be recruited from the Faculty of Health Sciences at Kahramanmaraş Sütçü Imam University and randomly assigned to one of the three groups using block randomization to ensure balanced allocation. All participants will initially receive a standardized 2-hour face-to-face theoretical session on Leopold maneuvers, delivered by experienced faculty members using the same content.

Following the theoretical instruction:

The video group will view a professionally prepared instructional video demonstrating all four Leopold maneuvers.

The model group will engage in hands-on practice using standardized pregnant anatomical mannequins under supervision.

The control group will not receive any additional material or practice after the theoretical session.

Psychomotor skill acquisition will be measured using a structured and validated 25-item Leopold Maneuver Psychomotor Skills Assessment Form, scored on a 0-4 Likert scale per item, with a total score range of 0-100. Assessments will be conducted at two time points: (1) within a few days following the intervention (to assess immediate skill gain), and (2) two months post-intervention (to assess skill retention).

To address potential ethical concerns and ensure educational equity, compensatory training (video + model-based) will be offered to all groups after final assessments are completed.

Additional data collection tools include:

A Student Satisfaction Scale designed for evaluating the learner experience with the instructional method,

The Spielberger State Anxiety Inventory (STAI-S) to assess state anxiety levels during skills application phases.

All statistical analyses will be conducted using SPSS version XX (or equivalent), employing appropriate tests for intergroup comparisons (e.g., ANOVA, repeated measures ANOVA) and within-group changes (e.g., paired t-tests or non-parametric equivalents depending on distribution). A p-value < 0.05 will be considered statistically significant.

The study adheres to ethical guidelines for human subject research and has obtained approval from the relevant Institutional Ethics Committee. Participation is voluntary and written informed consent will be obtained from all students prior to enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Must be a second-year student in the Department of Midwifery at -Kahramanmaraş Sütçü Imam University, Faculty of Health Sciences
* Has not previously taken the "Normal Pregnancy and Care" course
* Has not received prior training on Leopold maneuvers
* Willing to voluntarily participate in the study
* Able to attend all training and assessment sessions during the study period

Exclusion Criteria:

* Having an acute health condition that may interfere with participation in the training
* Being on leave or having frozen enrollment during the study period
* Sharing study content or violating confidentiality with members of other groups
* Withdrawing from the study voluntarily or being excluded due to absenteeism

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 99 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2025-11-15 (Estimated); Study Completion 2026-04-15 (Estimated)

PRIMARY OUTCOMES:
Psychomotor Skill Score in Leopold Maneuver Application | Assessed within 1 week after training and again at 8 weeks after training
  The primary outcome is the change in psychomotor skill scores measured by the Leopold Maneuver Psychomotor Skill Assessment Form. This validated tool consists of 25 observable items scored on a 5-point Likert scale (0-4), with a total score range of 0-100. Higher scores indicate greater proficiency in performing the Leopold maneuvers.

SECONDARY OUTCOMES:
Student Satisfaction with Training Method | Assessed within 1 week after training and again at 8 weeks after training
  Student satisfaction will be measured using a custom 6-point Likert scale ranging from 0 (not satisfied) to 5 (very satisfied), indicating the participant's perceived satisfaction with the instructional method used (video or model-based).
State Anxiety Level | Assessed within 1 week after training and again at 8 weeks after training
  Anxiety will be assessed using the Spielberger State Anxiety Inventory (SAI), which includes 20 items rated on a 4-point Likert scale. Scores range from 20 to 80, with higher scores indicating greater anxiety.

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared due to institutional policies and data privacy concerns.

REFERENCES:
- [Background] Opoku A, Usman MB, Adjei TA, Owusu-Afriyie B, Opoku W. Nursing and midwifery students' perceptions of sign language training in Ghana: relevance, instructional methods, and assessment practices. BMC Nurs. 2025 Jul 18;24(1):942. doi: 10.1186/s12912-025-03610-y. PMID 40682143
- [Background] Bowers M, Terry D, Irwin P. The impact of reflective practice on nursing students: a scoping review. Nurse Educ Pract. 2025 Aug;87:104468. doi: 10.1016/j.nepr.2025.104468. Epub 2025 Jul 13. PMID 40683080
- See also: Background This randomized controlled trial evaluated the outcomes of simulation- and video-based training for teaching nursing students Leopold's maneuver. Their self-efficacy and anxiety levels were also explored. Method Data were collected among 12 — https://journals.lww.com/simulationinhealthcare/abstract/2023/04000/evaluation_of_the_effectiveness_of_different.5.aspx